CLINICAL TRIAL: NCT00455585
Title: Comparison of the Steady State Pharmacokinetics of Nevirapine, Stavudine Plus Lamivudine in HIV Positive Ugandan Patients Taking Triomune 40 With the Pharmacokinetics of the Originator Products.
Brief Title: Comparison of Plasma Drug Levels of Triomune 40 With Those of the Originator Products
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Makerere University (Other)
Collaborators: Department of Foreign Affairs, Ireland (Other Government)
Responsible Party: Concepta Merry, Infectious Diseases Institute
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CPR001
Record Dates: First submitted 2007-04-02; First posted 2007-04-03 (Estimated); Last update posted 2008-02-08 (Estimated); Status verified 2008-02

CONDITIONS: HIV Infections
Keywords: Pharmacokinetics; Antiretrovirals; Uganda; HIV; Treatment Experienced
MeSH Terms: conditions — HIV Infections | interventions — stavudine, lamivudine, nevirapine drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: nevirapine, stavudine, lamivudine

SUMMARY:
This study aims to compare the steady state pharmacokinetics of stavudine, lamivudine, and nevirapine in HIV positive Ugandan patients taking Triomune 40 with the pharmacokinetics of the originator products known as Viramune, Epivir and Zerit 40.

DETAILED DESCRIPTION:
The introduction of combination antiretroviral therapy (ART) has revolutionised the treatment of HIV/AIDS. ART has been associated with significant reductions in morbidity and mortality mainly in wealthy countries and Brazil. ART which consists of a cocktail of at least three different potent anti-HIV drugs, has now been adopted as the standard of care for the management of HIV disease in developed countries.

The major constraint for widespread use of antiretrovirals (ARVs) in developing countries has been the high cost of drug acquisition and associated monitoring tests. The drug acquisition cost of innovator ARV ranges from €12,000 to €20,000 per patient per year. This compares with an annual cost of 558,000 Ugandan shilling or €260 per patient per year for Triomune, the most commonly generically manufactured ARV.

Triomune exists as two formulations, Triomune 40 and Triomune 30, both manufactured by Cipla Mumbai, India. Both contain nevirapine 200mg and lamivudine 150mg, however the Triomune 40 contains stavudine 40mg and Triomune 30 contains stavudine 30mg. This allows for the fact that persons weighing >60kg require a dose of stavudine 40mg and those weighing <60kg require a dose of stavudine 30mg. Therefore in patients weighing >60kg Tiomune 40 is prescribed, in patients <60kg Triomune 30 is prescribed. At the time of study design the majority of patients attending the Infectious Diseases Institute, Mulago Hospital and receiving ARV with Triomune were >60kg and therefore receiving Triomune 40.

The available pharmacokinetic data for Triomune is limited to a single dose study in healthy Indian volunteers which was performed by the manufacturer of Triomune, Cipla Mumbai and only one independent bioequivalence study on the steady state pharmacokinetic parameters of Triomune in HIV infected patients in Malawi. Of concern in this study Triomune was found not to be bioequivalent to the originator products with significantly higher d4T levels in the patients on Triomune when compared to the originator product. In this study the patients also reported more side-effects, principally peripheral neuropathy, when taking Triomune and the authors postulated that this may have been a result of the higher d4T levels in these patients. It was also noted that nevirapine levels were markedly higher in Malawians compared to western subjects of same weight, possibly due to genetic metabolic differences. The authors concluded that similar evaluation of drug exposure should be performed as these medications are introduced to new populations.

A study in the Cameroon examined the clinical outcome of 60 patients treated with Triomune over a 24 week period. This important study by Laurent et al. is the first published study addressing the issue of the quality of generic drugs and, as he points out, there are no clinical trials assessing the effectiveness, safety and quality of fixed dose combination drugs in resource limited environments. The study does however have several limitations. As the author himself acknowledges the sample size is small and therefore "not as powerful as a controlled trial". There is no comparison group taking branded (proprietary) drugs. The study time at 24 weeks is too short to satisfactorily assess the efficacy of these drugs- the European medicines Agency (EMEA), the European drug regulatory authority, requires a study period of 48 weeks for assessment of efficacy. Some major drug studies comparing different drug combinations have seen no significant difference in viral load suppression at 24 weeks but marked differences at 48 weeks. Laurent et al. performed in vitro dissolution testing on the drugs in their study; however this does not translate into bioequivalence. There are no bioequivalence data in this study. The authors did measure plasma trough drug levels at three time points as a measure of adherence but these measurements cannot be used to confirm bioequivalence.

Comparison(s) Steady state levels of stavudine, lamvivudine and nevirapine in HIV positive patients taking Triomune 40 for one month compared with the steady state levels of these agents when the originator products Zerit 40, Epivir and Viramune have been taken for one month, with patients acting as their own controls.

Pharmacogenomics

Pharmacogenomics is the study of the effect of genetic variation on drug disposition. It is a growing area of research and there is emerging data to support genomic differences in antiretroviral drug levels and related toxicity. There is increasing evidence that drug disposition varies between ethnic groups. In some cases this is due to different expression of the genes which encode the various components of the cytochrome system, in others it is felt to be linked to the varying expression of the genes encoding drug transporters. There is currently extremely limited data in this area relating to Africans. By storing blood samples from subjects enrolled in pharmacokinetic studies such as this a large and unique pharmacogenomic resource would be build up at Makerere University.

ELIGIBILITY:
Inclusion Criteria:

* Age over eighteen years Ability to provide full informed written consent Confirmed diagnosis of HIV infection On ARV therapy with Triomune 40

Exclusion Criteria:

* Haemoglobin < 8g/dl Liver and renal function tests > 3 times the upper limit of normal Pregnancy Use of know inhibitors or inducers of cytochrome P450 or P-glycoprotein. Use of herbal medications Weight <60kg Intercurrent illness

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18
Dates: Start 2007-01; Primary Completion 2007-05 (Actual); Study Completion 2007-11 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics of nevirapine, stavudine and lamivudine

SECONDARY OUTCOMES:
Safety aand tolerability of nevirapine, stavudine and lamivudine
Pharmacogenomics of Ugandan subjects

CONTACTS AND LOCATIONS:
Overall Officials: Concepta Merry, PhD, Principal Investigator — University of Dublin, Trinity College; Keith McAdam, Study Director — Infectious Diseases Institute, Makerere University
Locations (1):
- Makerere University, Infectious Diseases Insititute, Kampala, Uganda

REFERENCES:
- [Background] JA Gogtay, V.M., VG Nayak, PV Bodhe, A Dasgupta, V Srivatsan, G Vaidyanathan, KC Patel. A pharmacokinetic evaluation of lamivudine, stavudine and nevirapine given as a fixed dose combination pill versus the same three drugs given safely in healthy human volunteers. in 6th International Congress on Drug Therapy in HIV Infection. 2002. Glasgow,UK. 16.
- [Background] Laurent C, Kouanfack C, Koulla-Shiro S, Nkoue N, Bourgeois A, Calmy A, Lactuock B, Nzeusseu V, Mougnutou R, Peytavin G, Liegeois F, Nerrienet E, Tardy M, Peeters M, Andrieux-Meyer I, Zekeng L, Kazatchkine M, Mpoudi-Ngole E, Delaporte E. Effectiveness and safety of a generic fixed-dose combination of nevirapine, stavudine, and lamivudine in HIV-1-infected adults in Cameroon: open-label multicentre trial. Lancet. 2004 Jul 3-9;364(9428):29-34. doi: 10.1016/S0140-6736(04)16586-0. PMID 15234853
- [Background] Hosseinipour M C, C.A., Kanyama C, Mshali I. Pharmacokinetic Comparison of Generic and Trade Formulations of Lamivudine, Stavudine and Nevirapine in HIV-infected Malawian Subjects. in 12th Conference on Retroviruses and Opportunistic Infections. 2005. Boston. 17.